CLINICAL TRIAL: NCT07110844
Title: A Phase 2 Clinical Trial of Teclistamab and Daratumumab in Previously Untreated AL Amyloidosis
Brief Title: Teclistamab-Daratumumab in AL Amyloidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzanne Lentzsch, MD (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Suzanne Lentzsch, MD, Professor of Medicine and the Director of the Multiple Myeloma and Amyloidosis Program, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV8827; 1452862 (Other Grant/Funding Number: StandUp2Cancer (in collaboration with Janssen))
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Amyloid Light-chain Amyloidosis
Keywords: Untreated AL Amyloidosis; untreated light chain amyloidosis; light chain amyloidosis; AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Teclistamab-Daratumumab (Experimental): All participants in this study will receive teclistamab and daratumumab.
  Interventions: Drug: Teclistamab; Drug: Daratumumab and Hyaluronidase-fihj

INTERVENTIONS:
Drug: Teclistamab — Teclistamab is a T-cell redirecting bispecific antibody (BsAb) targeting CD3 on T-cells and B-cell maturation antigen (BCMA) on plasma cells.
  Other Names: TECVAYLI; teclistamab-cqyv
Drug: Daratumumab and Hyaluronidase-fihj — Daratumumab is an monoclonal antibody that targets the CD38 protein on the surface of myeloma cells.
  Other Names: DARZALEX FASPRO; Daratumumab

SUMMARY:
The purpose of this study is to investigate whether teclistamab-daratumumab combination is effective and safe in AL amyloidosis.

The study treatment is divided into cycles (C) and each cycle is 28 days (D). Study treatment is expected to last 6 months.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness and safety of teclistamab-daratumumab combination in newly diagnosed AL amyloidosis. The study aims to evaluate whether this combination is able to effectively decrease the level of toxic amyloid-producing light chains circulating in the participants' blood, with the overarching goal of avoiding organ damage, improving organ function, and prolonging life.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years and able to sign Informed Consent Form (ICF). If the individual being considered for participation in this study is unable to provide informed consent due to medical, cognitive, or other conditions, a legally authorized representative (LAR) may consent on their behalf.
2. Ability to comply with the study protocol, in the investigator's judgment.
3. Confirmed histopathological diagnosis of systemic AL amyloidosis by mass spectrometry or immunohistochemistry (IHC) or Immunofluorescence (IF) on a tissue biopsy that is positive for Congo Red.
4. Patient must not have received any prior plasma cell clone-directed therapy.
5. Measurable hematologic disease, defined as one of the following:

   1. Difference between involved and uninvolved serum free light chain (dFLC) ≥50 mg/L and/or 5 mg/dL
   2. Serum M-protein ≥0.5 g/dL on protein electrophoresis
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. One or more organs involved by AL amyloidosis as per consensus guidelines
8. Pre-treatment clinical laboratory values meeting the following criteria during the screening phase:

   1. Absolute neutrophil count ≥0.75 × 10^9/L
   2. Hemoglobin level ≥8.0 g/dL; red blood cell transfusion allowed until 7 days before C1D0.
   3. Platelet count ≥50 × 10^9/L; Platelet transfusions are acceptable without restriction during the Screening period
   4. Alanine aminotransferase level (ALT) ≤2.5 times the Upper Limit of Normal (ULN)
   5. Aspartate aminotransferase (AST) ≤2.5 times the ULN
   6. Total bilirubin level ≤1.5 × ULN except for subjects with Gilbert syndrome, in which case direct bilirubin ≤2 × ULN
   7. Estimated glomerular filtration rate (eGFR) ≥20 mL/min/1.73 m^2, measured by using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
9. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception and agreement to refrain from donating eggs.

For men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.

Exclusion Criteria:

1. Prior therapy for AL amyloidosis or multiple myeloma with the exception of 160 mg dexamethasone (or equivalent corticosteroid) maximum exposure prior to C1D0.
2. Patients meeting criteria for symptomatic multiple myeloma by any one of the following: (a) Lytic lesions on imaging (Skeletal survey, whole body CT or MRI, or PET/CT) (b) Plasmacytoma, (c) Hypercalcemia without any alternate etiology, (d) Bone marrow plasma cell infiltrate of greater than 60%.

   Patients with involved/uninvolved serum FLC ratio>100 as the sole myeloma-defining event will be allowed.
3. Evidence of significant cardiovascular conditions as specified below:

   1. NT-Pro BNP > 8500 pg/mL, and/or
   2. NYHA Class IIIb or IV functional class
4. History of other malignancy that could affect compliance with the protocol or interpretation of results.

   Patients with a history of curatively treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix, breast cancer, or Hodgkin's Lymphoma are generally eligible. Patients with a malignancy that has been treated, but not with curative intent, will be excluded, unless the malignancy has been in remission without treatment for ≥ 2 years prior to enrollment.
5. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal).
6. Patients on renal replacement therapy
7. Patients with HIV who are not on HAART or those with active hepatitis A, B, or C infection.
8. Planned stem cell transplant during the first 6 cycles of protocol therapy are excluded. Stem cell collection during the first 6 cycles of protocol therapy is permitted, as per investigators' discretion.
9. Known hypersensitivity to any of the agents
10. Patients who are receiving any other investigational agent concurrently.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Hematologic Complete Response (Heme-CR) rate | 6 months from treatment initiation
  Heme-CR will be defined as: involved free light-chain level less than the upper limit of the normal range with negative serum and urine immunofixation; normalization of the uninvolved free light-chain level or free light-chain ratio will not be required to determine a complete response.

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) negativity rate by Free Light Chain Mass Spectrometry (FLC-MS) in serum | 1 month, 3 months, 6 months, and 18 months
  Secondary outcome is to assess the rate of minimal residual disease (MRD)-negativity and sustained MRD-negativity with Teclistamab-Daratumumab
MRD-negativity rate by multiparameter flow cytometry (MFC) in bone marrow | 6 months and 18 months
  The MRD-negativity rate by 6 and 18 months will be reported descriptively.
Time to heme-CR | Day 1 of each cycle, and every 6 weeks after treatment cessation (up to 1 year)
  Time to heme-CR will be calculated from the day of treatment initiation (C1D0), and will be reported as median (range).
Major organ deterioration-progression-free survival (MOD-PFS) rate | From Cycle 2 to Cycle 6 Day 1 (Each cycle is 28 days), End of treatment visit (up to 6 months from treatment initiation), and up to 18 months from treatment initiation
  MOD-PFS will be calculated as a time-to-event endpoint using Kaplan-Meier method.
Overall survival rate | Through study completion, up to 18 months from treatment initiation
  Overall survival frequency from initiation of study drug, including cause of death for patients who die on study
Frequency of Cytokine Release Syndrome (CRS) | Throughout Cycle 1 (each cycle is 28 days), Day 0, Day 1, Day 3, Day 8, Day 15, Day 22; Throughout Cycle 2 and Cycle 6 on Day 1 and Day 15; End of treatment visit (up to 6 months from treatment initiation), Post treatment follow-up (up to 18 months)
  Frequency of CRS (all-grade and grade ≥3) events
Rate of infections | Throughout Cycle 1 (each cycle is 28 days), Day 0, Day 1, Day 3, Day 8, Day 15, Day 22; Throughout Cycle 2 and Cycle 6 on Day 1 and Day 15; End of treatment visit (up to 6 months from treatment initiation), Post treatment follow-up (up to 18 months)
  Frequency rate of infections (all-grade and grade ≥3) will be reported descriptively.
Number of participants with a heart response after treatment | 6 months and 18 months
  Heart response is defined as N-terminal pro Brain Natriuretic Peptide (NT-ProBNP) response (>30% and >300 ng/l decrease in subjects with baseline NT-proBNP>650 ng/l) or New York Heart Association (NYHA) class response (>2 class decrease in subjects with baseline NYHA class 3 or 4)
Number of No Responses in the heart after treatment | 6 months and 18 months
  No response in the heart is defined as ≤30% reduction in NT-proBNP from baseline
Number of Partial Responses (PR) in participants who experienced a heart response after treatment | 6 months and 18 months
  Partial Response in the heart is defined as 31-60% reduction in NT-proBNP from baseline.
Number of Very Good Partial Responses (VGPR) in participants who experienced a heart response after treatment | 6 months and 18 months
  VGPR in the heart is defined as >60% reduction in NT-proBNP from baseline to a nadir of >350 ng/L
Number of Complete Response (CR) in participants who experienced a heart response after treatment | 6 months and 18 months
  Complete Response in the heart is defined as Nadir NT-proBNP≤350 ng/L
Number of participants with heart progression after treatment | 6 months and 18 months
  Heart progression is defined as NT-proBNP progression (>30% and >300 ng/l increase) or cardiac troponin progression (>33% increase) or ejection fraction progression (>10% decrease). Subjects with progressive worsening renal function cannot be scored for NT-proBNP progression.
Number of participants with a kidney response after treatment | 6 months and 18 months
  Kidney response is defined as 50% decrease (at least 0.5 g/day) of 24-h urine protein (urine protein must be >0.5g/day pretreatment). Creatinine and creatinine clearance must not worsen by 25% over baseline.
Number of No Responses in the kidneys after treatment | 6 months and 18 months
  No response in the kidneys is defined as ≤30% reduction in proteinuria from baseline
Number of Partial Responses (PR) in participants who experienced a kidney response after treatment | 6 months and 18 months
  Partial Response in the kidneys is defined as 31-60% reduction in proteinuria from baseline
Number of Very Good Partial Responses (VGPR) in participants who experienced a kidney response after treatment | 6 months and 18 months
  VGPR in the kidneys is defined as >60% reduction in proteinuria from baseline level to a nadir level >200 mg/24 hours
Number of Complete Response (CR) in participants who experienced a kidney response after treatment | 6 months and 18 months
  Complete Response in the kidneys is defined as Nadir proteinuria ≤200 mg/24 hours
Number of participants with kidney progression after treatment | 6 months and 18 months
  Kidney progression is defined as 50% increase (at least 1 g/day) of 24-h urine protein to >1 g/day or 25% worsening of serum creatinine or creatinine clearance.
Number of participants with liver response after treatment | 6 months and 18 months
  Liver response is defined as 50% decrease in abnormal alkaline phosphatase value.
Number of No Responses in the liver after treatment | 6 months and 18 months
  No response in the liver is defined as ≤30% reduction in alkaline phosphatase (ALP) from baseline.
Number of Partial Responses (PR) in participants who experienced liver response after treatment | 6 months and 18 months
  Partial Response in the liver is defined as 31-60% reduction in ALP from baseline.
Number of Very Good Partial Responses (VGPR) in participants who experienced liver response after treatment | 6 months and 18 months
  VGPR in the liver is defined as >60% reduction in ALP from baseline to a nadir >2x lower limit of normal (LLN)
Number of Complete Response (CR) in participants who experienced liver response after treatment | 6 months and 18 months
  Complete Response in the liver is defined as Nadir ALP ≤2X LLN
Number of participants with liver progression after treatment | 6 months and 18 months
  Liver progression is defined as 50% increase of ALP from nadir value

OTHER OUTCOMES:
Hematologic event-free survival (Heme-EFS) | Throughout Cycle 2 and Cycle 6 (each cycle is 28 days) on Day 1; End of treatment visit (up to 6 months from treatment initiation), Post treatment follow-up (up to 18 months from treatment initiation)
  Heme-EFS will be calculated as a time-to-event endpoint using Kaplan-Meier method.
CD4 cell count | Baseline until 18 months from treatment initiation
  CD4 cells will be measured in participants before and after treatment.
CD8 cell count | Baseline until 18 months from treatment initiation
  CD8 cells will be measured in participants before and after treatment.
CD19 cell count | Baseline until 18 months from treatment initiation
  CD19 cells will be measured in participants before and after treatment.
IgG level | Baseline until 18 months from treatment initiation
  IgG titers will be measured in participants before and after treatment.
IgA level | Baseline until 18 months from treatment initiation
  IgA titers will be measured in participants before and after treatment.
IgM level | Baseline until 18 months from treatment initiation
  IgM titers will be measured in participants before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lentzsch, MD, PhD, Study Chair — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No